CLINICAL TRIAL: NCT03047460
Title: Feasibility and Reliability of Multimodal Evoked Potentials in an International Multicenter Setting
Status: Completed | Type: Observational
Sponsor: Clinique Neuro-Outaouais (Other)
Responsible Party: Principal Investigator, Dr. Francois Jacques, neurologist, Clinique Neuro-Outaouais
Other Study IDs: CNO-005
Record Dates: First submitted 2016-11-07; First posted 2017-02-09 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis
Keywords: motor evoked potential; somatosensory evoked potentials; biomarker
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy: healthy volunteers, 18 to 58 years old, with no neurological disease that could affect evoked potential responses
  Intervention: multimodal evoked potentials
  Interventions: Other: multimodal evoked potentials
- multiple sclerosis: All types of Multiple sclerosis patients:
  * Aged 18 to 58 years old, inclusive, at the time of informed consent.
  * Expanded Disability Status Scale (EDSS) 0.0 to 6.5.
  * Have measurable responses on both MEP and SSEP in at least one upper and one lower limb. The MEP and SSEP responses do not need to be in the same limb
  * Have no comorbid condition (ie neuropathy) that could affect testing.
  Intervention: multimodal evoked potentials
  Interventions: Other: multimodal evoked potentials

INTERVENTIONS:
Other: multimodal evoked potentials

SUMMARY:
Study Objectives and Endpoints:

Objective:

The primary objective of the study is to evaluate the feasibility and test-retest reliability of MEP's and (SSEP's) in a multicenter clinical trial in healthy subjects and subjects with MS.

Endpoints:

The primary reliability endpoint will be the intraclass correlation coefficient (ICC) of the following evoked potential parameters

DETAILED DESCRIPTION:
The establishment of a biomarker(s) that can predict a clinical response to therapy over the course of a 1-2 year clinical trial is critical for the expeditious development of treatments for Multiple Sclerosis (MS). Identification of this biomarker would enable shorter and smaller clinical trials resulting in the faster development of much needed treatments for MS, specifically neuro-reparative therapies. The etiology of disease progression is conduction block, demyelination and axonal degeneration. Evoked potentials provide a direct assessment of the underlying etiologies of disease progression in MS. They are a functional assessment of multiple pathways, including visual, motor and sensory, evaluating the integrity of myelin and axons.

The variability of motor evoked potentials (MEP) measures has limited multimodal evoked potential (mmEP) use in international, multicenter clinical trials. MEP evaluation does significantly contribute to the predictive value of mmEP's. Recent advances in technology and establishment of standardized protocols for MEP reduces the variability associated with this procedure. The objective of this study is to evaluate the reliability and feasibility of MEP and SSEP in an international, multicenter trial so that mmEP can be further evaluated as a biomarker for disease progression. The rationale for this study is to explore the feasibility and reliability of MEP's and somatosensory evoked potentials (SSEP's) in a multicenter clinical trial for potential use as a biomarker that can predict clinical progression/improvement in international clinical trials evaluating remyelinating therapies.

Study Objectives and Endpoints:

Objective:

The primary objective of the study is to evaluate the feasibility and test-retest reliability of MEP's and (SSEP's) in a multicenter clinical trial in healthy subjects and subjects with MS.

Endpoints:

The primary reliability endpoint will be the intraclass correlation coefficient (ICC) of the following evoked potential parameters

Motor Evoked parameters that will be measured:

* MEP latency
* Central motor conduction time (CMCT) root latency methods
* MEP amplitude
* MEP amplitude to compound motor amplitude ratio (MEP-M ratio) for the right and left abductor digiti minimi (ADM) and the right and left tibialis anterior (TA)
* Somatosensory evoked potential parameters will include Evoked potential latencies for both upper and lower limbs bilaterally.

Study Design:

This multinational, multicenter study will be conducted in healthy adult volunteers and MS patients to establish the feasibility and reliability of mmEP's. A total of 40 subjects, 10 (5 healthy and 5 MS) from each of the 4 sites will be enrolled.

The study will consist of two visits, 1-30 days apart, during which subjects will be screened to confirm eligibility and will complete all specified study assessments.

Study Locations:

Canada, Germany, Switzerland and Italy, with 1 site in each country.

Number of Planned Subjects:

A minimum of 40 subjects are planned for this study. Subjects who withdraw from the study prior to completion of the second visit may be replaced at the discretion of the investigator.

Study Population:

This study will be conducted in subjects 25 to 58 years of age, inclusive, who are either healthy volunteers (HV) or have been diagnosed with clinically definite MS who have a detectable lesion by MEP or SSEP.

Study Groups:

Two groups, healthy volunteers and clinically definite MS will be included.

Duration of Study Participation:

Study duration for each subject will be two visits, the second visit schedule >24 hours-30 days from the first visit

Criteria for Evaluation:

Key Study Assessments:

Electrophysiological. MEP's and SSEPs will be measured in both upper and lower limbs bilaterally. All studies will be read locally and reviewed by a blinded reader at another center. The ICC of every measured evoked potential parameter will be determined on both the central and local reads.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, candidates must meet the following eligibility criteria at Screening, or at the time point specified in the individual eligibility criterion listed (HV cohort):

  1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
  2. Aged 18 to 58 years old, inclusive, at the time of informed consent.
  3. Have no significant health issues, ie neuropathy or other demyelinating disorder that can affect testing.

Inclusion Criteria (MS Cohort)

To be eligible to be included in this cohort, candidates must meet the following additional eligibility criteria at Screening:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Aged 18 to 58 years old, inclusive, at the time of informed consent.
3. Diagnosis of MS (all types) with an expanded disability status scale (EDSS) 0.0 to 6.5.
4. Have measurable responses on both MEP and SSEP in at least one upper and one lower limb. The MEP and SSEP responses do not need to be in the same limb
5. Have no comorbid condition (ie neuropathy) that could affect testing.

Exclusion Criteria:

* Candidates will be excluded from study entry if any of the following exclusion criteria exist at screening or at any time during the study.

  1. Inability to comply with study requirements.
  2. Unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment.
  3. Any diseases (e.g., non-MS demyelinating diseases), with the exception of diagnosis MS for the MS Cohort, that in the opinion of the Investigator, could influence evoked potential results ( including but not limited to medullary trauma, morbid obesity, limb amputation, diabetes, other polyneuropathy).
  4. MS relapse within 3 months of either sessions.
  5. Initiation of treatment or dose adjustment within 1 month of either sessions with Fampyra, Tegretol, Baclofen, Zanaflex
  6. Febrile illness within 3 days of either sessions.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers and MS patients aged 18 to 58 that have no other neurological comorbities that could affect evoked potential responses
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Intraclass correlation coefficient (ICC) of the multi modal evoked potential parameters in order to determine the validity of the compound measures | obtained between two assessments done more than 24 hrs but less than 1 month apart
  multi modal evoked potential will include:
  * MEP latency (msec)
  * Central motor conduction time (CMCT) using root latency methods (msec)
  * MEP amplitude (mvolt) and MEP/CMAP amplitude ratio (%)

CONTACTS AND LOCATIONS:
Overall Officials: François Jacques, MD, Principal Investigator — Clinique Neuro-Outaouais
Locations (1):
- Clinique Neuro-Outaouais, Gatineau, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
the data will pooled with 3 other centers to augment the power of the study
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: for the duration of the study and completion of the analyses
Access Criteria: all PI's at each center will have access to the data